CLINICAL TRIAL: NCT01905436
Title: Optimization of Mass Drug Administration With Existing Drug Regimens for Lymphatic Filariasis and Onchocerciasis for Liberia
Brief Title: Mass Drug Administration for Lymphatic Filariasis and Onchocerciasis for Liberia
Acronym: DOLF-LIBERIA
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201107185
Record Dates: First submitted 2013-07-12; First posted 2013-07-23 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Lymphatic Filariasis; Onchocerciasis; Soil Transmitted Helminth (STH) Infections
Keywords: Filariasis; Onchocerciasis; Albendazole; Ivermectin; STH Soil Transmitted Helminth infections; MDA Mass Drug Administration
MeSH Terms: conditions — Elephantiasis, Filarial; Onchocerciasis; Infections; Filariasis | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Study procedures include collection of finger prick blood that will be tested for microfilaremia and for serology testing (antigenemia and antibody testing). Investigators will also collect skin snips (small superficial skin biopsies) to detect Onchocerca microfilariae, and stool samples to detect parasitic worm eggs indicative of STH infections.
  All assays will be performed in Liberia (filarial serology tests, MF smears, stool examinations).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Annual Mass Drug Administration: This group will receive annual mass drug administration (Albendazole 400 mg plus Ivermectin) provided by the Liberian Ministry of Health.
  Interventions: Drug: Annual versus Semiannual Albendazole plus Ivermectin Mass Drug Administration
- Semiannual Mass Drug Administration: This group will receive semi-annual mass drug administration (Albendazole 400 mg plus Ivermectin) provided by the Liberian Ministry of Health.
  Interventions: Drug: Annual versus Semiannual Albendazole plus Ivermectin Mass Drug Administration

INTERVENTIONS:
Drug: Annual versus Semiannual Albendazole plus Ivermectin Mass Drug Administration — Annual or semiannual Albendazole plus Ivermectin, administered by the Liberian Ministry of Health.
  Other Names: Albenza (Albendazole); Ivermectin, also known as Mectizan or Stromectol.

SUMMARY:
Approximately 5,200 people will participate per year. The study population will include females and males over 5 years of age who live in filariasis and onchocerciasis endemic areas. Subject selection will not be based on health status.

Two sites will be studied, and each study will last for 4 years. Participants will be studied only once in cross-sectional surveys. Some subjects may be included in more than one annual population survey, but this is not a longitudinal study.

Investigators will compare annual and semiannual mass drug administration (MDA) for lymphatic filariasis and onchocerciasis, and investigators will compare the impact of these MDA schedules on soil transmitted helminth infections. MDA will be administered by others (Liberian Ministry of Health or Liberian Institute of Biomedical Research).

The investigators will test the hypothesis that semiannual mass drug administration (MDA) is superior to annual MDA for elimination of lymphatic filariasis, onchocerciasis and for control of soil transmitted helminth (STH) infections.

1. Compare the relative impact and cost effectiveness of annual vs. twice yearly mass drug administration (MDA) for elimination of lymphatic filariasis (LF) in these populations.
2. Compare the relative impact and cost effectiveness of annual vs. twice yearly mass drug administration (MDA) for elimination of onchocerciasis in these populations.
3. Study the impact of annual vs. semiannual MDA on soil transmitted helminth (STH) infection in these populations.

Continuation Activities (2019/2020):

Additional one-time cross-sectional surveys will be completed in the Harper site in Maryland district in 2019 and in Lofa in 2020 to measure the long-term impact of MDA on W. bancrofti, O. volvulus, and on STH infection parameters following these cumulative 7-9 rounds of MDA since the baseline survey taken in 2013. Since the last DOLF surveys (3rd follow-ups) in these sites in 2016 & 2017, respectively, there have been a total of 3 annual rounds of MDA in both areas. These additional surveys will recruit 2,500 participants in the Maryland area villages and 3,200 in the Lofa area villages.

DETAILED DESCRIPTION:
Lymphatic filariasis (LF) is a deforming and disabling infectious disease that causes elephantiasis and genital deformity (especially hydroceles). The infection affects some 120 million people in 81 countries in tropical and subtropical regions with well over 1 billion people at risk of acquiring the disease [1]. LF is caused by Wuchereria bancrofti and Brugia spp. (B. malayi and B.timori), nematode parasites that are transmitted by mosquitoes. This study is based on the assumption that currently used MDA regimens and schedules are not optimal for achieving elimination of LF. These regimens (either annual Albendazole (Alb) 400 mg plus diethylcarbamazine 6 mg/kg or Alb 400 mg plus Ivermectin (Iver) 200 µg/kg for LF) were introduced more than 10 years ago.

Onchocerciasis ("Oncho") is similar in some ways to LF in that it is a vector-borne nematode parasitic disease that causes severe disability. In contrast to LF, this disease causes blindness and severe skin disease rather than elephantiasis, and it is spread by black flies instead of mosquitoes. O. volvulus adult worms live in subcutaneous nodules while the adult worms of the LF parasites live in lymphatic vessels. O. volvulus adult worms are larger and less sensitive to available drug treatments than those of the species that cause LF and have a longer lifespan (approximately 14 years rather than the estimated 7 years for LF parasites). More effective drugs or dosing schedules for MDA against Oncho could shorten the number of years needed to interrupt Oncho transmission in areas that previously had high disease rates.

Drugs used for LF MDA are also active against soil transmitted helminth infections (STH, e.g., Ascaris, Hookworm, and Trichuris). De-worming campaigns using anthelmintics usually target special groups of the population, such as schoolchildren, and have limited impact on transmission. Treatment of the total population and semiannual treatments may reduce re-infection considerably and will most likely lead to reduced infection densities and infection prevalence rates. Suppression of STH is an important ancillary benefit of MDA programs for filarial infections. Increasingly control programs for filariasis and STH are being integrated with programs for other parasitic diseases such as schistosomiasis. For this reason, participants will also be tested for schistosomiasis.

Purpose: The study aims to compare the effectiveness once yearly (1X) versus twice yearly (2X) mass drug administration (MDA) for the elimination of lymphatic filariasis, onchocerciasis and for control of soil-transmitted helminth infections (intestinal parasites) in large populations. Mass drug administration will be provided by the Liberian Ministry of Health. This project will assess the impact of the government's public health program.

Procedures: Study procedures include collection of finger prick blood that will be tested for microfilariae by microscopy and for serology testing (antigenemia and antibody testing). Skin snips will be collected and examined by microscopy for the presence of Onchocerca microfilariae. Stool samples will be collected for detection of parasitic worm eggs by microscopy. All assays will be performed in Liberia (filarial serology tests, microfilaria testing, stool examinations).

Washington University researchers developed the protocol, will provide training and guidance to Liberian researchers, and work with them to analyze the data. Liberian researchers will consent the participants, obtain blood, skin and stool specimens, perform laboratory tests on the specimens, and enter data on participants and lab results.

ELIGIBILITY:
Inclusion Criteria:

* • Study areas should be endemic for filariasis and onchocerciasis.
* • Study population have limited or no prior experience with MDA. Males and Females greater than 5 years of age.

Exclusion Criteria:

* • Children less than 5 years of age.
* • Children who weigh less than 15 kg (33 lb)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study populations are people who live in areas of Liberia that are co-endemic for lymphatic filariasis and onchocerciasis.
Sampling Method: Non-Probability Sample
Enrollment: 21862 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of W. bancrofti microfilaria (4 years) | 4 years
  Prevalence of W. bancrofti microfilaria (mf) is a binary outcome measured by the presence/absence of W. bancrofti mf in three-line thick smears prepared with a measured 60 microliter quantity of finger prick blood collected between 8pm-2am. The species of mf will be determined by morphological criteria.
Prevalence of W. bancrofti filarial antigenemia (4 years) | 4 years
  Prevalence of this outcome measure is determined by the percentage (%) of individuals with positive tests for the W. bancrofti filarial antigen. Blood will be tested for filarial antigenemia using the Alere Filariasis Test Strip (FTS).

SECONDARY OUTCOMES:
Prevalence of O. volvulus microfilaria (4 years) | 4 years
  Prevalence of O. volvulus microfilaria (mf) is a binary outcome measured by the presence/absence of O. volvulus mf taken from skin snips using Holth corneoscleral punches taken from the buttocks.
Community egg load of soil transmitted helminth (STH) eggs (4 years) | 4 years
  Community egg load is defined as average stool egg count per species. FLOTAC and Kato-Katz (KK) methods will be used to examine a single stool sample from each subject.
Prevalence of W. bancrofti microfilaria (7 years) | 7 years
  Prevalence of W. bancrofti microfilaria (mf) is a binary outcome measured by the presence/absence of W. bancrofti mf in three-line thick smears prepared with a measured 60 microliter quantity of finger prick blood collected between 8pm-2am. The species of mf will be determined by morphological criteria.
Prevalence of W. bancrofti filarial antigenemia (7 years) | 7 years
  Prevalence of this outcome measure is determined by the percentage (%) of individuals with positive tests for the W. bancrofti filarial antigen. Blood will be tested for filarial antigenemia using the Alere Filariasis Test Strip (FTS).
Prevalence of O. volvulus microfilaria (7 years) | 7 years
  Prevalence of O. volvulus microfilaria (mf) is a binary outcome measured by the presence/absence of O. volvulus mf taken from skin snips using Holth corneoscleral punches taken from the buttocks.
Community egg load of soil transmitted helminth (STH) eggs (7 years) | 7 years
  Community egg load is defined as average stool egg count per species. FLOTAC and Kato-Katz (KK) methods will be used to examine a single stool sample from each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Weil, MD, Principal Investigator — Washington University School of Medicine; Peter U Fischer, PhD, Principal Investigator — Washington University School of Medicine; Fatorma K Bolay, PhD, Study Director — Liberian Institute of Biomedical Research
Locations (1):
- Liberian Institute of Biomedical Research, Charlesville, Margibi County, Liberia

REFERENCES:
- See also: Death to Onchocerciasis and Lymphatic Filariasis (DOLF) Project — http://www.dolf.wustl.edu/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT01905436/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT01905436/ICF_001.pdf